CLINICAL TRIAL: NCT00159120
Title: Maintenance Treatment vs. Stepwise Drug Discontinuation After One Year of Maintenance Treatment in First-Episode Schizophrenia
Brief Title: Maintenance Treatment vs. Stepwise Drug Discontinuation in First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network On Schizophrenia (Network); Janssen-Cilag Ltd. (Industry); University of Bonn (Other); Humboldt-Universität zu Berlin (Other); Ludwig-Maximilians - University of Munich (Other); University of Göttingen (Other); University of Cologne (Other); Mainz University (Other); University Hospital Tuebingen (Other); Universität Duisburg-Essen (Other); University of Mannheim (Other); University of Jena (Other); Martin-Luther-Universität Halle-Wittenberg (Other); RWTH Aachen University (Other); University of Wuerzburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01GI 9932 - P 2.2.2.1 / 2
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia; Psychoses
Keywords: Schizophrenia; first episode; neuroleptic maintenance treatment; drug discontinuation; prodrome based early intervention
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): further maintenance antipsychotic treatment and prodrome-based early intervention
  Interventions: Other: maintained antipsychotic treatment vs. stepwise drug discontinuation
- 2 (Experimental): stepwise drug discontinuation (after 1 year maintenance antipsychotic treatment) and prodrome-based early intervention
  Interventions: Other: maintained antipsychotic treatment vs. stepwise drug discontinuation

INTERVENTIONS:
Other: maintained antipsychotic treatment vs. stepwise drug discontinuation — maintained antipsychotic treatment (in low dose) vs. stepwise drug discontinuation; both supplemented by prodrome-based early intervention; 1 year

SUMMARY:
After one year neuroleptic maintenance treatment in patients with first episode schizophrenia, neuroleptic treatment will be continued vs. stepwise discontinued (randomized design) over a period of 1 year. Under both conditions prodrome based early intervention take place.

DETAILED DESCRIPTION:
After one year neuroleptic maintenance treatment in patients with first episode schizophrenia, neuroleptic treatment will be continued vs. stepwise discontinued (randomized design) over a period of 1 year. Under both conditions pharmacologic early intervention strategies in case of early sign of relapse will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients after 1 year of maintenance treatment after their first-episode in schizophrenia (according ICD-10 F20)
* Age between 18 and 55
* Informed consent
* One year neuroleptic maintenance treatment
* Reaching stable course

Exclusion Criteria:

* Residence outside of the catchment area
* Legal reasons
* Insufficient knowledge of the german language
* Substance abuse or addiction
* Pregnancy
* Serious physical illness
* Organic brain disease
* Contraindication to neuroleptic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2001-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
relapse rate | 1 year

SECONDARY OUTCOMES:
psychopathology | 1 year
social and cognitive functioning | 1 year
side-effects | 1 year
drop-out | 1 year
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Gaebel, Professor, Study Chair — Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University of Düsseldorf, Rhineland State Clinics Düsseldorf, Bergische Landstraße 2, 40629 Düsseldorf, Germany
Locations (1):
- German Research Network on Schizophrenia, Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Gaebel W, Moller HJ, Buchkremer G, Ohmann C, Riesbeck M, Wolwer W, Von Wilmsdorff M, Bottlender R, Klingberg S. Pharmacological long-term treatment strategies in first episode schizophrenia--study design and preliminary results of an ongoing RCT within the German Research Network on Schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2004 Apr;254(2):129-40. doi: 10.1007/s00406-004-0509-y. PMID 15146342
- [Derived] Seemuller F, Schennach R, Mayr A, Musil R, Jager M, Maier W, Klingenberg S, Heuser I, Klosterkotter J, Gastpar M, Schmitt A, Schlosser R, Schneider F, Ohmann C, Lewitzka U, Gaebel W, Moller HJ, Riedel M; German Study Group on First-Episode Schizophrenia. Akathisia and suicidal ideation in first-episode schizophrenia. J Clin Psychopharmacol. 2012 Oct;32(5):694-8. doi: 10.1097/JCP.0b013e3182677958. PMID 22926606
- [Derived] Gaebel W, Riesbeck M, Wolwer W, Klimke A, Eickhoff M, von Wilmsdorff M, Lemke M, Heuser I, Maier W, Huff W, Schmitt A, Sauer H, Riedel M, Klingberg S, Kopcke W, Ohmann C, Moller HJ; German Study Group on First-Episode Schizophrenia. Relapse prevention in first-episode schizophrenia--maintenance vs intermittent drug treatment with prodrome-based early intervention: results of a randomized controlled trial within the German Research Network on Schizophrenia. J Clin Psychiatry. 2011 Feb;72(2):205-18. doi: 10.4088/JCP.09m05459yel. Epub 2010 Jun 29. PMID 20673559
- See also: Click here for more information about this study: Pharmacological long-term treatment strategies for relapse prevention in first episode schizophrenia — http://www.kompetenznetz-schizophrenie.de